CLINICAL TRIAL: NCT02181582
Title: Evaluation of Specific PET Radioligand Binding To Translocator Protein
Brief Title: Specific PET Radioligand Binding to Translocator Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 140141; 14-M-0141
Record Dates: First submitted 2014-07-02; First posted 2014-07-04 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2016-11-23

CONDITIONS: Baseline; Blocking Receptor Binding
Keywords: Health Humans; Receptor Occupancy

ARMS (1):
- Emapunil Administration (Experimental): Single Arm Study
  Interventions: Drug: Emapunil; Device: PET

INTERVENTIONS:
Drug: Emapunil — Single peroral administration
Device: PET — Positron emission tomography, which creates images by detecting radioactivity.

SUMMARY:
Background:

- A brain protein called translocator protein (TSPO) shows changes in some brain diseases. A radioactive drug called 11C-(R)-PK 11195 is used to take pictures of TSPO using a camera called positron emission tomography (PET). Researchers want to find out how well 11C-(R)-PK 11195 takes the pictures.

Objective:

- To evaluate the radioactive chemical 11C-(R)-PK 11195.

Eligibility:

- Healthy volunteers ages 18-55.

Design:

* Participants will be screened with a medical exam.
* Participants will have scans at up to 4 visits.

  * PET scan using 11C-(R)-PK 11195:

    * A small tube (catheter) will be put into an artery at the wrist or elbow, by a needle. The needle will be removed, leaving only the catheter in the artery. Blood samples will be taken through this catheter.
    * Another catheter will be placed into a vein in the arm or hand.
    * 11C-(R)-PK 11195 will be injected through the second catheter.
    * The PET scanner is shaped like a doughnut. Participants will lie on a bed that slides in and out of it. They may get a plastic mask for their face and head.
  * Participants will receive a dose of emapunil by mouth. Participants will then have another PET scan.
  * Participants may have a magnetic resonance imaging (MRI) scan. The MRI scanner is a metal cylinder surrounded by a magnetic field. The participant will lie on a table that can slide in and out of the cylinder. Participants will get earplugs for the loud knocking noises.
* After each scan, participants will get a follow-up phone call. Two to seven days after taking emapunil, participants will return for a follow-up visit.

DETAILED DESCRIPTION:
Objective:

The 18kDa Translocator Protein (TSPO, formerly known as the peripheral benzodiazepine receptor (PBR)) is expressed in activated microglia and reactive astrocyte. It has therefore been used as an imaging target for positron emission tomography (PET) to investigate diseases involving microglial activation and/or macrophage recruitment, such as multiple sclerosis, herpes encephalitis, Parkinson s disease, Alzheimer s disease and ischemic stroke. The vast majority of PET studies reported to date have used 11C-(R,S) and 11C-(R)-PK 11195, a 3-isoquinolinecarboxamide antagonist, with nanomolar affinity for TSPO. Several second generation radioligands, including 11C-PBR28, 11C-DPA-713, and 11C-ER176 have been developed. Although these ligands have greater signal to noise (specific to nondisplaceable uptake) ratio than 11C-(R)-PK 11195,their binding to TSPO is affected by a single nucleotide polymorphism (SNP). Specific to nondisplaceable ratio of 11C-PBR28 has recently been reported. However, no one has ever measured the specific to nondisplaceable ratio of other TSPO radioligands including 11C-(R)-PK 11195, 11C-DPA-713 and 11C-ER176 in human subjects. In addition, differences in this binding site between species preclude comparisons based on studies in animals. The purposes of this study are to measure the signal to noise ratio (i.e., ratio of specific to non-displaceable uptake) of 11C-(R)-PK 11195, 11C-ER176 and 11C-DPA-713 in human subjects with two scans in each subject: at baseline and after emapunil, an agonist at the TSPO site and a putative anxiolytic based on studies in animals and in humans and study the effect of the SNP on the in vivo specific binding of the PET ligands.

Study population:

75 healthy volunteers in total aged 18 to 55 years. Of these, 25 will have 11C-(R)-PK 11195, 25 have 11C-DPA-713 scans, and 25 have 11C-ER176.

Design:

Healthy volunteers (n = up to 25) will have two scanning sessions using 11C-(R)-PK 11195: a) baseline i.e., medication-free and b) blocking i.e. with medication. For blocking, we will give one oral dose of emapunil (15 or 90 mg), about 1.5 hours before the second injection of the radioligand. Both scanning sessions would include an arterial line and measurement of the input function of parent radioligand separated from radiometabolites as well as plasma free fraction of radioligand. Additional 25 healthy volunteers will have two scanning sessions using 11C-DPA-713 in the same design, one baseline and another after one oral dose of emapunil. An additional 25 healthy volunteers will have two scanning sessions using 11C-ER176 in the same design, one baseline and another after one oral dose of emapunil. The total number of participants is 75 (= 25 + 25 + 25)

Outcome measures:

Baseline scans measure total binding i.e., total distribution volume (V[T]). By applying the Lassen plot, combined data from both baseline scans and those with administration of emapunil measure nonspecific binding i.e., nondisplaceable distribution volume (V[ND]). From these V[T] and V[ND] values, specific-to-nondisplaceable ratios will be calculated as (V[T] V[ND]) / V[ND[ and the influence of the SNP to specific binding, V[S] = V[T] - VND will also be studied.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Male or female subjects between 18 to 55 yrs of age and able to give written informed consent.
  2. Subjects must be healthy based on medical history, physical examination and laboratory testing.
  3. Be able to provide own consent.
  4. Agree to use contraception for 30 days after emapunil administration.

EXCLUSION CRITERIA:

1. Any past or present Axis I psychiatric disorder. Any history of alcohol or substance dependence, except nicotine dependence, within the past 6 months
2. Serious medical problems including but not limited to chronic neurological disease such as multiple sclerosis, autoimmune diseases, or serious cardiopulmonary disease.
3. Active seizure disorder, as defined as having had a seizure in the past year or being on antiepileptic medications for seizures.
4. Positive HIV test.
5. Recent research-related exposure to radiation (i.e., PET from other research) which when combined with this study would be above the allowable limits.
6. Metallic foreign bodies that would be affected by the MRI magnet or fear of enclosed spaces likely to make the subject unable to undergo an MRI scan.
7. Claustrophobia
8. Positive urine drug screen at time of enrollment.
9. Pregnancy at time of scan (beta-HCG will be measured in all female patients within 24 hours before start of scan and must be negative). Lactating women who are breast feeding.
10. Prescription or over-the counter medication use; psychotropic herb use (e.g., St. John s Wort).
11. Are not able to comfortably lie flat on the back for at least two and a half hours at a time

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-24; Primary Completion 2016-06-16 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
Signal noise ratio [C-11](R)-PK 11195 | 2 moths

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Fujita, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States